CLINICAL TRIAL: NCT04140994
Title: Effects of rTMS on Brain Plasticity and Motor Learning in Healthy People.
Brief Title: Innovative Brain Stimulation for Induction of Learning Plasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Pierre Nicolo, Principal Investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Project-ID 2019-01440 CCER
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent theta burst stimulation (Active Comparator): Volunteers will be submitted to non-invasive parietal stimulation before a mirror drawing task.
  A transcranial magnetic stimulator (MagPro X100, Medtronic Functional Diagnostics, Skovlunde, Denmark) will deliver interrmittent bursts of bipolar magnetic pulses exerting an excitation on the underlying brain tissue (iTBS). The stimulation coil will be placed over the parietal cortex. Stimulation consisted of a burst of three pulses administered at 50Hz, repeated at a frequency of 5Hz, delivered in 2 s trains followed by an 8 s interval for a total of 600 pulses12. Stimulation intensity was set at 70% of RMT.
  Each session will consist of two spaced neuronavigated iTBS applications, separated by 15 minutes.
  Interventions: Device: rTMS device
- Sham intermittent theta burst stimulation (Sham Comparator): For sham iTBS, the protocol is the same, except the sham coil produces no magnetic field.
  Interventions: Device: rTMS device

INTERVENTIONS:
Device: rTMS device — Participants will participate in 1 session of neuronavigated (TMS Navigator, Localite, Schloss Birlinghoven, D-53757, Sankt Augustin, Germany ) iTBS (patterned form of TMS) coupled with motor learning.

SUMMARY:
Recent studies have identified new neurobiological biomarker (i.e. functional connectivity of the parietal cortex) of motor learning among healthy people. This enables to refine our current model of motor learning wherein specific cortical processes are key factors for motor acquisition. Furthermore, recent evidence suggests that new technical approaches such as repetitive magnetic stimulation (rTMS) can efficiently influence this key factor. However, up to now, no rTMS studies have target this new biomarker. Therefore, the effect of rTMS are unknown. Hence, the investigators want to develop a new rTMS setup able to induce specific brain processes in healthy individuals that are likely to benefit. This has the potential to obtain critical information in order to improve treatment of motor re-learning in patients with neurological diseases.

DETAILED DESCRIPTION:
Participants will participate in 1 session of neuronavigated (TMS Navigator, Localite, Schloss Birlinghoven, D-53757, Sankt Augustin, Germany ) iTBS (patterned form of rTMS) coupled with motor learning. Participants will be randomly assigned to one of 2 groups: real iTBS over parietal cortex and sham iTBS over the parietal cortex.

One day before (Day1) and after the motor learning (Day 2), participants will undergo high-density 128-channel resting state electroencephalography (EEG) and motor evoked potential (MEP) in order to characterize the effects of rTMS on our markers of plasticity. Performance on the task will be measure immediately after learning (Day 2) and again 24h later (Day 3) in order to test for retention and offline consolidation (time and errors). The task will consist in realizing a computerized mirror-drawing task, in which right-left movements of the mouse were reversed on the screen.

ELIGIBILITY:
Inclusion Criteria:

* man or woman aged between 18-40 years,
* ability to give informed consent,
* ability to follow protocol instructions,
* normal or corrected-to-normal vision,

Exclusion Criteria:

* history of epileptic seizure (ci. TMS),
* skull breach (ci. TMS),
* metallic object in the brain (ci. TMS),
* pacemaker (ci. TMS),
* severe co-morbidity (ex, traumatic, rheumatologic, neurodegenerative diseases),
* pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Motor performance in consolidation test | after training (Day 3)
  Difference in error rate and speed improvement in active and sham groups (learned task)

SECONDARY OUTCOMES:
Resting state EEG connectivity in active and sham groups | Before (Day 1) and after training (Day 2)
  Calculated from electroencephalography recordings
Motor Evoked Potential (MEPs) Amplitudes (peak to peak) | Before (Day 1) and after training (Day 2)
  Difference in MEPs between active and sham groups. MEPs are generated when stimulation of the brain on the motor cortex (with Transcranial Magnetic Stimulation [TMS]) causes the spinal cord and peripheral muscles to produce neuroelectrical signals. MEPs are typically measured in the hand muscles (Abductor pollicis brevis ).

OTHER OUTCOMES:
Motor performance in retention test | After training (Day 2)
  Difference in error rate and speed improvement in active and sham groups (learned task)
Motor performance in transfer test | after training (Day 2 and Day 3)
  Difference in error rate and speed improvement in active and sham groups (non-learned) task)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Guggisberg, Prof. Dr., Study Director — University Hospital, Geneva
Locations (1):
- Pierre Nicolo, Geneva, Switzerland